CLINICAL TRIAL: NCT06527794
Title: Remote Hypertension Tracking, Help, and Management to Reduce Disparities in Black Patients
Brief Title: Remote Hypertension Management for Black Patients
Acronym: RHYTHM-B
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00112245; BPS-2023C1-31377 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Uncontrolled Hypertension
Keywords: high blood pressure; African-American population; remote blood pressure monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RHYTHM (Remote Hypertension Tracking Help Management) (Experimental): home blood pressure telemonitoring with remote medication management and social support, lifestyle education and connection to community resources to address social needs
  Interventions: Behavioral: RHYTHM (Remote Hypertension Tracking Help Management)
- Enhanced usual care (UC) (Experimental): standardized packet with evidence-based hypertension education material and a blood pressure monitor to complete blood pressure measurements at home
  Interventions: Behavioral: Enhanced usual care (UC)

INTERVENTIONS:
Behavioral: RHYTHM (Remote Hypertension Tracking Help Management) — Home blood pressure telemonitoring with remote medication management by a centralized multidisciplinary team led by a pharmacist; and social support, lifestyle education and connection to community resources to address social needs, provided by a community health worker who is embedded with the centralized team and is tightly connected to community resources and partners
  Arms: RHYTHM (Remote Hypertension Tracking Help Management)
Behavioral: Enhanced usual care (UC) — All participating sites will receive training on appropriate blood pressure measurement and education on guideline-based hypertension therapy. Additionally, participants in usual care will receive a standardized packet with evidence-based hypertension education material and a blood pressure monitor to complete blood pressure measurements at home.
  Arms: Enhanced usual care (UC)

SUMMARY:
This study will compare two approaches for managing hypertension in Black patients with uncontrolled blood pressure (BP). One approach will include home BP telemonitoring supported by a pharmacist and a community health worker. The other approach will include usual clinic-based care along with a home BP monitor and routine care.

DETAILED DESCRIPTION:
This study is a pragmatic effectiveness-implementation hybrid type 2 trial with two study arms. One arm will include home BP telemonitoring supported by a pharmacist and a community health worker providing centralized self-management support. The other arm will include enhanced usual clinic-based care with a home BP monitor and routine care from providers trained on evidence-based guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Black or African American race
* Hypertension diagnosis
* aged 21 to 85 years
* Uncontrolled blood pressure as defined by [a] most recent SBP ≥140 mmHg and an additional SBP≥140 mmHg within the past 12 months in an outpatient setting (excluding urgent care, emergency department or surgery clinic), or [b] most recent SBP>160mmHg in an outpatient setting (excluding urgent care, emergency department or surgery clinic), or [c] referral by PCP for uncontrolled hypertension with at least one documented SBP≥140 mmHg (in clinic or at home) in the past 12 months; and (v) primary care provided at a participating clinic.
* Able to speak English
* Primary care provided at a participating clinic

Exclusion Criteria:

* currently pregnant or planning to get pregnant during the study period
* residence in a long-term care facility, hospice or with a terminal illness with less than 1 year life expectancy as determined by the Primary Care Physician or study team. Stable chronic illness such as compensated cirrhosis, chronic obstructive pulmonary disease, congestive heart failure etc. will not be excluded.
* estimated Glomerular Filtration Rate (eGFR) <30 ml/min or on dialysis. Patients with a functioning kidney transplant will not be excluded.
* inability to provide informed consent or participate in study procedures. For example, conditions that limit ability to participate in phone visits or check BPs in at least one arm.
* currently participating in another BP management program.
* plan to move out of the area within the next 12 months.
* Hispanic ethnicity.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Blood pressure control - Percent of patients achieving BP control (i.e., Systolic BP<130mmHg) - Month 12 | Month 12
  Percent of patients achieving BP control (i.e., SBP<130mmHg)

SECONDARY OUTCOMES:
Blood pressure control - Percent of patients achieving BP control (i.e., Systolic BP<130mmHg) - Baseline | Baseline
  Percent of patients achieving BP control (i.e., SBP<130mmHg)
Blood pressure control - Percent of patients achieving BP control (i.e., Systolic BP<130mmHg) - Month 6 | Month 6
  Percent of patients achieving BP control (i.e., SBP<130mmHg)
Blood pressure control - Percent of patients achieving BP control (i.e., Systolic BP<130mmHg) - Month 18 | Month 18
  Percent of patients achieving BP control (i.e., SBP<130mmHg)
Systolic blood pressure (mmHg) - Baseline | Baseline
  Mean SBP (mmHg)
Systolic blood pressure (mmHg) - Month 6 | Month 6
  Mean SBP (mmHg)
Systolic blood pressure (mmHg) - Month 12 | Month 12
  Mean SBP (mmHg)
Systolic blood pressure (mmHg) - Month 18 | Month 18
  Mean SBP (mmHg)
Self-Management - Hypertension Self-Care Profile Score - Baseline | Baseline
  The hypertension self-care profile score encompassed self-care behaviors crucial to control blood pressure - Includes 3 scales (Behavior, Motivation, Self-efficacy) 20 items each that can be used together or independently. The Behavior scale assesses participant's self-care behaviors on a 4-point Likert scale. Mean scores range from 1-4 with higher scores indicating higher levels of self-care behavior. The Motivation scale assesses participant's self-care motivation on a 4-point Likert scale. Mean scores range from 1-4 with higher scores indicating higher levels of self-care motivation. The Self-efficacy scale assesses participant's self-care efficacy on a 4-point Likert scale. Mean scores range from 1-4 with higher scores indicating higher levels of self-efficacy. Higher scores indicate better self care behaviors - range from 60-240.
Self-Management - Hypertension Self-Care Profile Score - Month 12 | Month 12
  The hypertension self-care profile score encompassed self-care behaviors crucial to control blood pressure - Includes 3 scales (Behavior, Motivation, Self-efficacy) 20 items each that can be used together or independently. The Behavior scale assesses participant's self-care behaviors on a 4-point Likert scale. Mean scores range from 1-4 with higher scores indicating higher levels of self-care behavior. The Motivation scale assesses participant's self-care motivation on a 4-point Likert scale. Mean scores range from 1-4 with higher scores indicating higher levels of self-care motivation. The Self-efficacy scale assesses participant's self-care efficacy on a 4-point Likert scale. Mean scores range from 1-4 with higher scores indicating higher levels of self-efficacy. Higher scores indicate better self care behaviors - range from 60-240.
Medication adherence - Hill-Bone medication adherence scale survey score - Baseline | Baseline
  Hill-Bone medication adherence scale survey - 14-item Hill-Bone Compliance Scale uses a 4-point Likert scale. Score range from 14-56. Higher scores indicates poorer adherence.
Medication adherence - Hill-Bone medication adherence scale survey score - Month 12 | Month 12
  Hill-Bone medication adherence scale survey - 14-item Hill-Bone Compliance Scale uses a 4-point Likert scale. Score range from 14-56. Higher scores indicates poorer adherence.
Patient assessment of chronic illness care (PACIC) survey score - Baseline | Baseline
  The Patient assessment of chronic illness care (PACIC) survey assess implementation of the chronic care model from the patient perspective. The PACIC includes five subscales addressing specific domains: (1) patient activation; (2) delivery system design/decision support; (3) goal setting/tailoring; (4) problem solving/contextual counselling; and (5) follow-up/coordination. Patients rated care received from their healthcare team (e.g., physicians, nurses, physiotherapists, occupational therapists, social workers) during the past 6-months using a 5-point Likert scale (1 = 'never' to 5 = 'always'). Total and subscale scores (i.e., summed items completed within that scale) are averaged across items.
Patient assessment of chronic illness care (PACIC) survey score - Month 12 | Month 12
  The Patient assessment of chronic illness care (PACIC) survey assess implementation of the chronic care model from the patient perspective. The PACIC includes five subscales addressing specific domains: (1) patient activation; (2) delivery system design/decision support; (3) goal setting/tailoring; (4) problem solving/contextual counselling; and (5) follow-up/coordination. Patients rated care received from their healthcare team (e.g., physicians, nurses, physiotherapists, occupational therapists, social workers) during the past 6-months using a 5-point Likert scale (1 = 'never' to 5 = 'always'). Total and subscale scores (i.e., summed items completed within that scale) are averaged across items.
20-Item Short Form Health Survey (SF-20) - Baseline | Baseline
  The SF-36 Total/Global/Overall Score, a global measure of health-related quality of life - scores range from 0-100 with higher scores denoting better quality of life
20-Item Short Form Health Survey (SF-20) - Month 12 | Month 12
  The SF-36 Total/Global/Overall Score, a global measure of health-related quality of life - scores range from 0-100 with higher scores denoting better quality of life
Healthcare Utilization - Number of Acute Care Days - Baseline | Baseline
  Total days spent in an emergency department, inpatient hospital, or observation unit; number of physician office visits.
Healthcare Utilization - Number of Acute Care Days - Month 12 | Month 12
  Total days spent in an emergency department, inpatient hospital, or observation unit; number of physician office visits.
Healthcare Utilization - Number of Acute Care Days - Month 24 | Month 24
  Total days spent in an emergency department, inpatient hospital, or observation unit; number of physician office visits.

OTHER OUTCOMES:
Therapeutic intensification Score | Month 12
  The therapeutic intensity score is a number that reflects the number of medications and the percent of maximal dose of each medication. Numeric range 0-5.

CONTACTS AND LOCATIONS:
Overall Officials: Yhenneko J. Taylor, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Patient-Centered Outcomes Research Institute (PCORI) Data Management and Data Sharing Policy, will prepare a Full Data Package (analyzable data set, full protocol, metadata, data dictionary, full statistical analysis plan and analytic code) for access by third parties. Per PCORI policy, the Full Data Package will be maintained at Atrium Health for 7 years, unless required by PCORI to be deposited in a separate repository.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The Policy calls for maintenance of the Full Data Package for seven (7) years following acceptance by PCORI of the Final Research Report. In that time, PCORI may provide funds for the deposition of the Full Data Package to the PCORI-designated repository in circumstances where PCORI requests such deposition (e.g., due to PCORI estimate of high importance of research project findings or external research request).
Access Criteria: Individual investigators or teams of investigators seeking access to data from PCORI-funded studies must complete and submit a data request form to the PCORI-designated repository. There are no categorical restrictions on what types of individuals or entities may request to access the PCORI Awardee research data. Data requestors will be evaluated for their overall qualifications and experience (e.g., across a proposed team of specified individuals) to achieve the stated research purpose underlying the data request.